CLINICAL TRIAL: NCT04404179
Title: Setting up a COVID-19 Care Facility at a Prison in Pakistan
Status: Completed | Type: Observational
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Usman Ismat Butt, Assistant Professor, Services Institute of Medical Sciences, Pakistan
Other Study IDs: CovJ
Record Dates: First submitted 2020-05-24; First posted 2020-05-27 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19; Prison; Pakistan
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CASE: 59 COVID-19 POSITIVE PRISONERS WHO UNDERWENT TREATMENT AT THE COVID-19 CARE FACILITY AT CAMP JAIL.
  Interventions: Other: COVID-19 FACILITY

INTERVENTIONS:
Other: COVID-19 FACILITY — A COVID-19 facility was setup within the Prison. All positive prisoners were managed in the facility. If further intervention was required they were to be shifted to Services Hospital , Lahore.

SUMMARY:
Presenting outline of the steps taken by our team to set up a Covid Care facility within the Prison setting. The facility was set up at Camp Jail (Lahore District Jail) located on Ferozpur Road, Lahore.

DETAILED DESCRIPTION:
A prisoner brought to Camp Jail developed symptoms of and later tested positive for COVID-19. This lead to almost 527 contacts. An outbreak was expected. To manage the situation , a COVID-19 Care Facility was established within the prison. The study describes the steps taken by the team to set up this facility.

ELIGIBILITY:
Inclusion Criteria:

- All COVID-19 positive prisoners within the Camp Jail

Exclusion Criteria:

* Any patient being shifted to any other facility (except designated)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population consisted of the prisoners who after being exposed to a suspected COVID-19 patient tested positive on screening. a total of 59 prisoners were detected by screening. They were included in the study. 10 COVID-19 prisoners shifted to Camp Jail were also latter included.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Recovery | 30 days
  Confirmed by double negative PCR results of specimen obtained via nasopharyngeal swabs
Mortality | 30 days
  Death of any of the patients who had tested positive at the Camp Jail
ICU admission | 30 days
  Any patient requiring admission to intensive care unit due to developing symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Camp Jail / COVID-19 CARE FACILITY/ SIMS, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No